CLINICAL TRIAL: NCT05589493
Title: Hybrid Polyetheretherketone (PEEK)-Acrylic Resin Prostheses and the All-on-4 Concept for Full-Arch Rehabilitation - Routine Group
Brief Title: Hybrid PEEK-Acrylic Resin Prostheses and the All-on-4 Concept for Full-Arch Rehabilitation - Routine Group
Acronym: AO4PEEKRG
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Malo Clinic (Other)
Collaborators: Invibio Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AO4PEEKRoutGroup
Record Dates: First submitted 2022-10-18; First posted 2022-10-21 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2022-10

CONDITIONS: Prosthesis Survival
Keywords: prosthesis; PEEK; All-on-4; All-on-four; dental implants
MeSH Terms: conditions — Prosthesis Failure

STUDY DESIGN:
Intervention Model Description: Prospective cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All-on-4 PEEK routine (Experimental): Prosthetic full-arch rehabilitation using a PEEK-acrylic resin prosthesis
  Interventions: Device: Prosthetic full-arch rehabilitation using a PEEK-acrylic resin prosthesis

INTERVENTIONS:
Device: Prosthetic full-arch rehabilitation using a PEEK-acrylic resin prosthesis — A prosthetic full-arch rehabilitation of atrophic maxillae using a PEEk-acrylic resin prosthesis supported by dental implants following the All-on-4 Concept arrangement.
  Other Names: PEEK prosthesis

SUMMARY:
The goal of this observational study is to evaluate the outcome of a Poly-ether-ether-ketone - acrylic resin prosthesis for full-arch rehabilitation of the atrophic maxillae through the All-on-4 concept after five years of follow-up. The main question it aims to answer is:

- What is the survival outcome of the full-arch implant-supported Poly-ether-ether-ketone - acrylic resin prosthesis? The participants already rehabilitated with dental implants will receive a Poly-ether-ehter-ketone prosthesis as a definitive prosthesis.

DETAILED DESCRIPTION:
Following the learning generated during a development study with implant supported fixed prostheses using polyetheretherketone (PEEK) material, it is necessary to evaluate the outcome of implant supported fixed prosthetic rehabilitations using PEEK material in a routine scenario, following optimized laboratory and treatment protocol.

The study design will be a prospective single cohort to evaluate the long term outcome of fixed prosthetic implant supported rehabilitations. The cohort will be evaluated at 6 months, 12 months and annually thereafter until 5 years of follow-up. At each follow-up assessments multiple evaluaitons will be performed to assess the overall outcome of the restorations.

ELIGIBILITY:
Inclusion Criteria:

* Patients rehabilitated with immediate function implants for complete edentulous arches through the All-on-4 Concept.
* Patients in need of definitive implant-supported restorations.
* Written informed consent from each patient to participate in the study.

Exclusion Criteria:

- Hindrance to provide written informed consent. (A patient cannot participate if no written consent is given)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2017-11-13 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Survival of the prosthesis | 5 years
  Evaluation of the survival for the PEEK-acrylic resin implant-supported prosthesis; nominal (survival,failure)

SECONDARY OUTCOMES:
Survival of the implants | 5 years
  Evaluation of the survival for implants supporting the PEEK-acrylic resin implant-supported prosthesis; nominal (survival,failure)
Incidence of biological complications | 5 years
  Peri-implant infection, abscess, fistulae, suppuration, sinus infection, gingival dehiscence; Nominal (no incidence, incidence)
Incidence of mechanical complications | 5 years
  Loosening or fracture of prosthetic components; Nominal (no incidence, incidence)
Marginal bone resorption | 5 years
  Measured through periapical radiographs, in mm between the implant shoulder and the most apical portion of implant-bone contact; Scale
Denture staining | 5 years
  Veneer discoloration or staining. If JUVORA is exposed same discoloration or staining 0:heavily stained; 10: no stains
In mouth comfort | 5 years
  Visual analogue scale (0-10 cm); 0:very poor; 10: very good
Overall chewing feeling | 5 years
  Visual analogue scale (0-10 cm); 0:very poor; 10: very good
Oral Health Impact Profile OHIP-14 | 5 years
  Likert Scale (0=least impact/never, 4=highest impact/very often)
Patient tissue reaction | 5 years
  Visual analogue scale (0-10 cm); 0:very poor; 10: very good
Framework integrity | 5 years
  Visual analogue scale (0-10 cm); 0:very poor; 10: very good
Veneer adhesion | 5 years
  Visual analogue scale (0-10 cm); 0:very poor; 10: very good
Manufacture issues | 5 years
  Visual analogue scale (0-10 cm); 0:very poor; 10: very good
Handling of material compared to metal | 5 years
  Visual analogue scale (0-10 cm); 0:very poor; 10: very good
Aesthetics | 5 years
  Visual analogue scale (0-10 cm); 0:very poor; 10: very good
Speech | 5 years
  Visual analogue scale (0-10 cm); 0:very poor; 10: very good
Fit | 5 years
  Visual analogue scale (0-10 cm); 0:very poor; 10: very good
Hygiene around the implants | 5 years
  Visual analogue scale (0-10 cm); 0:very poor; 10: very good
Hygiene - how much plaque/calculus adheres to the prosthesis | 5 years
  Visual analogue scale (0-10 cm); 0:very poor; 10: very good
Overall classification from KOL | 5 years
  Visual analogue scale (0-10 cm); 0:very poor; 10: very good

CONTACTS AND LOCATIONS:
Overall Officials: Miguel A de Araújo Nobre, PhD, Principal Investigator — Director of Research, Development and Education
Locations (1):
- Malo Clinic, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: Yes
Anonymized database containing the study variables
Supporting Information: SAP
Time Frame: Upon study completion and for 8 years.
Access Criteria: Upon solicitation to the Investigators